CLINICAL TRIAL: NCT03128008
Title: Phase II Study of Accelerated and Adaptive Radiation Therapy for Locally-Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Locally Advanced NSCLC Hyperfractionated RT
Acronym: ADAPT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00083154
Record Dates: First submitted 2017-04-18; First posted 2017-04-25 (Actual); Results first posted 2020-02-24 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Carcinoma, Non Small Cell Lung (NSCLC)
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Carboplatin/Paclitaxel with radiation therapy (Experimental): Single arm, non randomized, open label study. Eligible subjects will receive standard of care Carboplatin IV once a week, Paclitaxel IV once a week given concurrently with daily hyperfractionated radiation therapy (RT). RT will be delivered as 6 fractions weekly.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Radiation: Daily hyperfractionated radiation therapy

INTERVENTIONS:
Drug: Carboplatin — Single arm non randomized open label study. Subjects will receive standard of care Carboplatin IV once a week. Chemotherapy is given concurrently with daily hyperfractioned radiation therapy.
Drug: Paclitaxel — Single arm non randomized open label study. Subjects will receive standard of care Paclitaxel IV once a week. Chemotherapy is given concurrently with daily hyperfractioned radiation therapy.
Radiation: Daily hyperfractionated radiation therapy — All subjects will receive 6 fractions(2Gy per fraction) of radiation therapy weekly. All subjects will complete an interim PET-CT after 48Gy-54Gy of RT . Subjects with a complete response on PET will complete RT at 60 Gy; subjects who have residual disease on interim PET and meet strict planning constraints eligibility will proceed to boost RT for a total RT dose of 72Gy. Interim PET-CT response will be measured using PERCIST criteria.

SUMMARY:
This is a prospective phase II study designed to evaluate an accelerated and adaptive RT approach for locally-advanced non-small cell lung cancer (NSCLC). All eligible subjects will have an interim PET-CT during radiation therapy to determine the metabolic complete response rate. Radiation therapy will be given in an accelerated fashion (2 Gy/fraction, 6 fractions/week) with concurrent chemotherapy. Interim responses will be assessed using PERCIST criteria.

Despite concurrent chemotherapy and radiation therapy, local/regional failure occurs in ~50% of patients with locally-advanced NSCLC. Clinical studies have demonstrated that accelerated fractionation (giving the same total dose in a shorter period of time) improves outcomes in several malignancies, including lung cancer. Administering higher than conventional doses of RT to all sites of original disease leads to inferior outcomes. Adapting the RT approach, giving a higher dose to slowly responding disease as assessed with interim PET has been shown to be feasible. PERCIST (Positron Emission Tomography Response Criteria in Solid Tumors) provides guidelines on how to report responses to therapy based on PET-CT. PET-CT response has been shown to be prognostic in a variety of clinical scenarios in lung cancer including after induction therapy. In one study, PET was performed after neoadjuvant chemoradiotherapy (40-50.4 Gy). Complete or partial metabolic response using PERCIST criteria was predictive of loco-regional, distant, and overall progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic/cytologic documentation of non-small cell lung cancer (NSCLC)
2. Unresectable stage II, IIIA, or IIIB disease
3. Zubrod/ECOG performance status 0-1
4. Weight loss < 10% in preceding 3 months prior to diagnosis
5. Adequate organ function defined as the following
6. Absolute neutrophil count of ≥ 1,500 and platelet count ≥ 100,000
7. Cockcroft calculated creatinine clearance of ≥ 45 ml/min or 1.5 x the upper limit of normal (ULN)
8. A total bilirubin ≤ 1.5 ULN, aspartate aminotransferase (AST) ≤ 2.0 x ULN
9. ≥ 18 years of age.
10. Negative pregnancy test in women of child-bearing potential
11. Signed study-specific informed consent.
12. No prior chemotherapy or radiotherapy for NSCLC
13. No prior mediastinal or thoracic radiation

Exclusion Criteria:

1. Prior thoracic irradiation.
2. Medical contraindications to thoracic irradiation.
3. Pre-existing sensory neuropathy of grade ≥ 2
4. Pleural effusion: when pleural fluid is visible on both CT scan and on a chest x-ray, a pleuracentesis is required to confirm that the pleural fluid is cytologically negative.

   Patients with effusions that are minimal (i.e. not visible on chest x-ray) or that are too small to safely tap are eligible
5. Patients with contralateral hilar involvement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2019-01-16 (Actual); Study Completion 2021-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kelsey, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Carboplatin/Paclitaxel With Radiation Therapy: Eligible subjects will receive standard of care Carboplatin IV once a week, Paclitaxel IV once a week given concurrently with daily hyperfractionated radiation therapy (RT). RT will be delivered as 6 fractions weekly.
Period: Overall Study
Arm/Group | Carboplatin/Paclitaxel With Radiation Therapy
Started | 10
Completed | 1 (9 participants are in follow up)
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Carboplatin/Paclitaxel With Radiation Therapy
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (7.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: The Metabolic Complete Response Rate, Assessed Using Interim PET-CT, in an Accelerated Fashion (2 Gy/Fraction, 6 Fractions/Week) With Concurrent Chemotherapy
Description: For the cohort of the participants who meet eligibility criteria and receive radiotherapy with concurrent chemotherapy, the metabolic complete response (MCR) rate will be measured with interim PET-CT utilizing PERCIST response reporting criteria.
Time Frame: 4 weeks
Population: 8 participants have RECIST measurements available
Measure: Count of Participants; unit: Participants
Groups:
- Carboplatin/Paclitaxel With Radiation Therapy: Eligible participants will receive standard of care Carboplatin IV once a week, Paclitaxel IV once a week given concurrently with daily hyperfractionated radiation therapy (RT). RT will be delivered as 6 fractions weekly.
Arm/Group | Carboplatin/Paclitaxel With Radiation Therapy
Number analyzed (Participants) | 8
Participants
  Progressive Disease | 1
  Stable Disease | 6
  Partial Response | 1
  Complete Response | 0

2. Secondary Outcome: The Number of Participants Eligible for an RT Boost After Completing a Standard Dose of RT (60 Gy), Delivered in an Accelerated Fashion (6 Fractions/Week) With Concurrent Chemotherapy
Description: In the same participant cohort, the proportion of the participants who are eligible for an RT boost after completing a standard dose of RT (60 Gy), delivered in an accelerated fashion (6 fractions/week) with concurrent chemotherapy, will be estimated as well as its confidence interval.
Time Frame: 4 weeks
Population: 9 participants indicated whether they had Boost or not
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin/Paclitaxel With Radiation Therapy
Number analyzed (Participants) | 9
Participants | 3

3. Secondary Outcome: Overall Survival With an Accelerated and Adaptive RT Approach.
Description: The overall survival (OS) for the treated participants will be characterized by Kaplan-Meier estimator. The medial OS will be estimated with a 95% confidence interval.
Time Frame: 2 years
Population: 1 participant did not have any follow up data
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carboplatin/Paclitaxel With Radiation Therapy
Number analyzed (Participants) | 9
months | NA [NA to NA] — The median survival time was not estimable due to the small sample size (2 in 9 participants were deceased). It was not possible to calculate the lower 95% confidence interval because the median survival (50% patients deceased in the cohort) was not reached.

4. Secondary Outcome: Progression-free Survival (PFS) With an Accelerated and Adaptive RT Approach.
Description: Median progression-free survival for participants will be characterized by Kaplan-Meier estimator. The median PFS will be estimated as well as their 95% confidence intervals.
Time Frame: 2 years
Population: One participant did not have any follow up data
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carboplatin/Paclitaxel With Radiation Therapy
Number analyzed (Participants) | 9
months | 13.39 [2.58 to NA] — The upper confidence level could not be measured due to the small sample size.

5. Secondary Outcome: Number of Participants With Local Control With an Accelerated and Adaptive RT Approach
Description: The local control rate for the same cohort of participants will be measured by standard of care imaging per NCCN guidelines at routine follow up clinic visits.
Time Frame: 2 years
Population: One participant does not have any follow up data.
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin/Paclitaxel With Radiation Therapy
Number analyzed (Participants) | 9
Participants | 1

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Carboplatin/Paclitaxel With Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 2/10
Serious Adverse Events (participants affected / at risk) | 6/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin/Paclitaxel With Radiation Therapy (N=10)
Allergic reaction (Immune system disorders) | 2
Esophageal Ulcer (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Cardiac troponin T increased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin/Paclitaxel With Radiation Therapy (N=10)
Anemia (Blood and lymphatic system disorders) | 3 (7)
Lymphocyte count decreased (Investigations) | 8 (17)
Neutrophil Count decreased (Investigations) | 6 (9)
White blood cell decreased (Investigations) | 7 (13)
Aspartate aminotransferase increased (Investigations) | 2 (4)
Weight loss (Investigations) | 8 (10)
Palpitations (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 4 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 5 (9)
Vomiting (Gastrointestinal disorders) | 3 (4)
Fatigue (General disorders) | 9 (11)
Non-cardiac chest pain (General disorders) | 3 (3)
Pain (General disorders) | 3 (4)
Mucosal infection (Infections and infestations) | 2 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 7 (10)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 4 (5)
Glucose intolerance (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 5 (6)
Anxiety (Psychiatric disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
cardiac disorders -other specify (Cardiac disorders) | 1 (1)
chest pain, cardiac (Cardiac disorders) | 1 (1)
esophageal ulcer (Gastrointestinal disorders) | 1 (1)
esophagitis (Gastrointestinal disorders) | 8 (9)
Fever (General disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 5 (5)
Papulopustular rash (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
alanine aminotransferase increased (Investigations) | 3 (3)
alkaline phosphatase increased (Investigations) | 1 (2)
lymphocyte count increased (Investigations) | 1 (1)
platelet count decreased (Investigations) | 1 (1)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
hypertension (Vascular disorders) | 1 (1)
hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/08/NCT03128008/Prot_SAP_000.pdf